CLINICAL TRIAL: NCT06505915
Title: Carbohydrate Loading Fasting Protocol Versus 'Sip Til Send': A Randomised Trial of Two Different Fasting Protocols at Elective Caesarean Delivery
Brief Title: Carbohydrate Loading Fasting Protocol Versus 'Sip Til Send'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Rotunda Hospital (Other)
Responsible Party: Principal Investigator, Rana Muhammad Shoaib Sadiq, Anaesthesia Fellow, The Rotunda Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: REC-2023-026
Record Dates: First submitted 2024-06-30; First posted 2024-07-17 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Elective Cesarean Delivery; Fasting ( 6H for Solid ; 2H for Clear Fluid )
Keywords: cesarean section and fasting protocols
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group C (Experimental): fasting protocol consuming carbohydrate drinks before elective caesarean delivery and sipping water until called to theatre
  Interventions: Dietary Supplement: Pre op Carbohydrate drink
- Group S (Active Comparator): fasting protocol NOT consuming carbohydrate drinks before elective caesarean delivery, but encouraged to sip water until called to theatre
  Interventions: Other: Clear fluid as per sip til send policy

INTERVENTIONS:
Dietary Supplement: Pre op Carbohydrate drink — Lemon flavoured clear carbohydrate drink
  Arms: Group C
Other: Clear fluid as per sip til send policy — clear fluid such as water
  Arms: Group S

SUMMARY:
Women undergoing elective caesarean deliveries are fasted for long periods prior to surgery. Recently, Rotunda Maternity Hospital have started using two fasting protocols at the Rotunda prior to elective caesarean section, one uses carbohydrate drinks, and the other encourages women to sip water until they are called to the operating theatre. The evidence to support the use of either one is very limited. This study would help streamline one of the protocols.

DETAILED DESCRIPTION:
This is a study focused on comparing fasting policies that are in use at the Rotunda.

Investigators wish to determine the best fasting policy for women at elective caesarean delivery by focusing on assessing outcomes related to the patient experience.

A 'Sip til send' fasting policy means women may drink clear fluid up until the time they are called from the ward to come to theatre for their elective caesarean delivery. This policy was implemented at the Rotunda in 2022 and was studied prospectively, investigators demonstrated improvements in the comfort that women experience in their perioperative journey, compared to a traditional fasting protocol where women must fast for many hours for both fluids and solids before they come to theatre.

It has been shown that oral carbohydrate intake may improve outcomes in general and cardiac surgeries, but there is very limited evidence in obstetrics. The Rotunda is increasingly providing women with carbohydrate drinks prior to CD. These drinks are consumed by the patient on the morning of surgery as part of an enhanced recovery after surgery (ERAS) package. There is little evidence to support the use of carbohydrate drinks, but current thinking is that they may increase energy and comfort and reduce metabolic changes due to prolonged fasting.

Pregnant women are more vulnerable to the side effects related to the extended fasting due to the accelerated fasting in the third trimester of pregnancy after an overnight fast pre-operatively. Carbohydrate reserves are rapidly exhausted, causing hypoglycemia, increased urine nitrogen secretion (indicating muscle catabolism), and increased urinary ketone body concentration. It has been recommended that Mothers in their third trimester avoid skipping meals.

Investigators wish to study the effects of integrating carbohydrate drinks into the current 'sip til send' fasting protocol and determine if these women benefit from either protocol.

ELIGIBILITY:
Inclusion Criteria:

* Elective caesarean section for singleton pregnancy under neuraxial anaesthesia.
* Subjects able to give informed consent and willing to comply with the study protocol.
* Subjects must be greater than 18 years old

Exclusion Criteria:

* Diabetes Mellitus - including gestational diabetes.
* Known foetal abnormality.
* Planned general anaesthesia.
* Elective caesarean delivery at a gestation of less than 37 weeks.
* Low birth weight 2.5 kg (IUGR)
* BMI greater than 45 kg/m2
* Women with severe gastro-oesophageal reflux disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All pregnant patients coming in for elective caesarean sections
Enrollment: 100 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
General well-being of the patient | Immediately Preoperatively
  Compare fasting protocols using a 0-10 Visual Analogue Score (VAS) for patient-focused comfort outcomes, including anxiety, thirst, hunger, nausea, and comfort. Each of them would be scored from 0 to 10, 0 being nothing and 10 being the maximum score relative to the feeling

SECONDARY OUTCOMES:
General well-being of the patient | 24 hours post operative
  1. Intraoperative nausea and vomiting: Assessed as YES or NO
  2. Pre-operative urinary ketone level: Assessed with urine dipstick showing POSITIVE or NEGATIVE
  3. Pre-operative blood sugar level: Measured on glucometer in mmol/lt
  4. Quality of recovery score following ceaserean delivery (ObsQoR11) score at 24 hours: consists of 11 questions related to how the symptoms have been in the last 24 hours regarding pain, vomiting, dizziness, shivering, comfort level, mobility, and the requirement of assistance related to looking after one's self and the baby. Each aspect is measured from a scale of 0 to 10, 0 being minimal and 10 being maximum.

CONTACTS AND LOCATIONS:
Locations (1):
- Rotunda Maternity Hospital, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sadiq RS, Murphy C, Drew T. A carbohydrate loading fasting protocol versus 'Sip til Send': a randomised trial of two different fasting protocols at elective caesarean delivery. BMC Anesthesiol. 2025 Oct 14;25(1):495. doi: 10.1186/s12871-025-03340-3. PMID 41087945